CLINICAL TRIAL: NCT04124562
Title: Nitrous Oxide Frequency of Use and Causes in Hospital in Turkey
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hilmi Demirkiran, MD, Department of Anesthesiology and Reanimation, Yuzuncu Yil University
Other Study IDs: Nitrous oxide
Record Dates: First submitted 2019-10-08; First posted 2019-10-11 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Environmental-Pollution-Related Condition
Keywords: Nitrous oxide; Prevalence; Turkey
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nitrous Oxide — Nitrous Oxide use ratio in Turkey's hospitals

SUMMARY:
The prevalence of nitrous oxide use in hospitals in Turkey

DETAILED DESCRIPTION:
Nitrous oxide has a long history of use in the healthcare field for over 150 years. However, this gas is slowly being abandoned for various reasons. The decrease in N2O use is probably due to its side effects and negative impact on global warming. Proven side effects include irreversible toxic effects on bone marrow, relative or absolute contraindications related to neuro and cardiac anesthesia, increased incidence of post-operative nausea and vomiting, increased risk of miscarriage in pregnant women (5), the greenhouse effect of nitrous oxide. In 2013, B. Husum et al. investigated the frequency of N2O use in public hospitals in Scandinavian countries and it was confirmed that N2O use was reduced and limited. According to the results of this research, N2O was administered with a volatile anesthetic agent in 21.5% of general anesthesia applications in Scandinavian countries. N2O was used as the second agent in Denmark by 2.4%, Finland by 17%, Iceland by 34.5, Norway by 32.1%, Sweden by 27.5%. In Turkey there are not enough reports of N2O use prevalence. In this study, we will investigate the extent of use and avoidance reasons N2O in Turkey. And we aim creating awareness.

ELIGIBILITY:
Inclusion Criteria:

Hospitals who accept to participate in Turkey

-

Exclusion Criteria:

Hospitals refusing to participate in the study

Age Groups: Child, Adult, Older Adult
Study Population: Anesthesiologists working in the operating rooms of hospitals in Turkey
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
The percentage of nitrogen oxide use | A day
  Percentage of nitrogen oxide use in a daily general anesthesia practice

SECONDARY OUTCOMES:
The percentage of nitrogen oxide use | A month
  Percentage of nitrogen oxide use in a monthly general anesthesia practice

CONTACTS AND LOCATIONS:
Overall Officials: Hilmi Demirkıran, 1, Principal Investigator — Study Director
Locations (1):
- Yuzuncu Yil University, School of Medicine, Van, Tusba / Zeve Kampus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No